CLINICAL TRIAL: NCT01963897
Title: Duchenne Muscular Dystrophy in Norway. Genotype/Phenotype in Patients Younger Than 18 Years, With a Main Focus on Growth, Puberty, Bone Health and Quality of Life.
Brief Title: Duchenne Muscular Dystrophy < 18y in Norway: Genotype/Phenotype, Growth, Puberty, Bone Health and Quality of Life.
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: The Research Council of Norway (Other); University Hospital of North Norway (Other)
Responsible Party: Principal Investigator, Magnhild Rasmussen, Dr.med., Oslo University Hospital
Other Study IDs: 2013/513
Record Dates: First submitted 2013-10-12; First posted 2013-10-16 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Genotype/phenotype correlations; Growth; Bone health; Puberty; Quality of life
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — whole blood, serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The study will give a consent based epidemiological overview of Norwegian patients with Duchenne muscular dystrophy younger than 18 years of age. Genotype of the population will be described. Longitudinal development of growth, bone health, and , when applicable, puberty over a two year period will be studied. Questionnaires regarding quality of life will also be an important part of the study.

DETAILED DESCRIPTION:
The participants who are not regularly seen at our regional hospital, are recruited via their local neuropediatrician. Patients who do not come to our region hospital will be seen at their local hospital.Each participant will be seen up to three times with one year between each visit. The visits include clinical examination, DXA scan, x-ray for bone age, and blood tests including several parameters related to bone health, growth and puberty. Standardized questionnaires regarding quality of life (patients and parents) will be used, and certain questions regarding the importance of achieving normal height and puberty will be added. Additional anamnestic data will be retrieved from the patients' medical records.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Duchenne muscular dystrophy
* Age under 18 years
* Residing in Norway

Exclusion Criteria:

-

Max Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients with Duchenne muscular dystrophy under 18 years in Norway
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2013-08; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Genotype | 1 day (At first visit)
  Specific description of mutation

CONTACTS AND LOCATIONS:
Overall Officials: Magnhild Rasmussen, Dr.med., Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No